CLINICAL TRIAL: NCT06120764
Title: Effect of Guided Imagery on Chemotherapy-related Nausea and Vomiting in Pediatric Oncology Patients: a Randomized Controlled Trial
Brief Title: Effect of Guided Imagery on Chemotherapy-related Nausea and Vomiting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe Ay, RN, PhD, Assistant Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KA23/180
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-02

CONDITIONS: Chemotherapy-induced Nausea and Vomiting; Pediatric Cancer
MeSH Terms: conditions — Vomiting; Neoplasms | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Intervention Model Description: The children in the experimental group will listen to the "Guided Imagery CD" prepared by the Turkish Psychological Association for relaxation 30 minutes before the chemotherapy infusion started and during the chemotherapy infusion. In the meantime, patients will be encouraged to think of various images, such as imagining that the treatment is over, returning to their old life quickly, etc.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be randomly assigned to groups. An independent statistician will analyze the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided imagery group (Experimental): Participants will receive guided imagery intervention.
  Interventions: Other: guided imagery
- Control (No Intervention): Participants will receive routine care.

INTERVENTIONS:
Other: guided imagery — The children in the experimental group will listen to the first part of the 'Guided Imagery CD' prepared by the Turkish Psychological Association for relaxation 30 minutes before the chemotherapy infusion starts. The suggestions given in the first part of the CD will help the patients relax and focus their attention on their breathing. Patients will be positioned in a supine or semi-fowler position and will listen to the CD with headphones from a laptop. Once the chemotherapy infusion starts, relaxing light background music with the sound of a river or sea will be played based on the patients' preference, and imagery will be applied to the patients. Patients will be encouraged to think of various images, such as imagining that the treatment is over, visualizing themselves as much healthier and recovering quickly, returning to their old life, and doing whatever they want to do first after recovery. If there is an object, person, event, situation, or food that will make them feel good,
  Arms: Guided imagery group

SUMMARY:
The goal of this randomized controlled study is to assess the effect of guided imagery on chemotherapy-related nausea and vomiting in pediatric oncology patients.

Participants will receive either guided imagery+routine care or routine care. The researchers will compare nausea and vomiting and vital signs between groups.

DETAILED DESCRIPTION:
Despite significant advances in anti-emetic treatment, chemotherapy induced nausea and vomiting (CINV) is considered a major side-effect that significantly reduces the quality of life of children diagnosed with cancer. Guided imagery is one of the methods of distraction that allows the individual to go to an environment or scene that will make the individual comfortable, peaceful, happy, and focused. In this study, the participants will be randomized in a single blind manner (participant) to either intervention or control groups.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 18 years old,
* who will receive intravenous chemotherapy,
* no cognitive or neurological disease that would prevent communication,
* receiving a chemotherapy protocol with a high or moderate emetogenic effect according to the MASCC/ESMO Antiemetic Guideline Classification,
* no verbal, visual and auditory communication disabilities (ability to speak Turkish, no mental deficiency),
* children whose parents and themselves volunteered to participate in the study

Exclusion Criteria:

* Children receiving radiotherapy,
* taking ginger powder or vitamins to reduce nausea,
* children who did not want to participate in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Nausea and vomiting | 30 minutes before the procedure, halfway through the chemotherapy infusion, immediately after the procedure, and for the first 24 hours after the end of chemotherapy
  Nausea and Vomiting Thermometer Scale in Children with Cancer is a 5-likert type scale. An increase in the score indicates an increase in the degree of nausea and vomiting experienced by children with cancer.

SECONDARY OUTCOMES:
Heart rate | 30 minutes before the procedure, halfway through the chemotherapy infusion, and immediately after the procedure,
  Maintaining or normalizing heart rate within normal range (60 to 110 bpm)
Systolic and diastolic blood pressure | 30 minutes before the procedure, halfway through the chemotherapy infusion, and immediately after the procedure
  Maintaining or normalizing systolic and blood pressure within normal range (systolic: 90-120 mmHg; diastolic 60-80 mmHg)
Respiratory rate | 30 minutes before the procedure, halfway through the chemotherapy infusion, and immediately after the procedure
  Maintaining or normalizing respiratory rate within normal range (18-30 breath per minute)
Body temperature | 30 minutes before the procedure, halfway through the chemotherapy infusion, and immediately after the procedure
  Maintaining or normalizing body temperature within normal range (36-37 C° in tympanic measurement)
Oxygen saturation | change from baseline 60 minutes of chemotherapy infusion
  Maintaining or normalizing oxygen saturation within normal range (between 95%-100% by pulse oximetry)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Ay, RN, PhD, Principal Investigator — Baskent University
Locations (1):
- Hacettepe University İhsan Doğramacı Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
the data wil be shared upon a reasonable request.